CLINICAL TRIAL: NCT04297306
Title: The Use of Virtual Reality Exercise Games to Improve Prehabilitation Exercise Compliance in Patients Awaiting Bariatric Surgery
Brief Title: Virtual Reality Exercise Gaming in Patients Awaiting Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020.RCHT.08
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Bariatric Surgery; Prehabilitation

STUDY DESIGN:
Intervention Model Description: Case-controlled trial randomised, prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise prescription (Active Comparator): This group will be provided with a prescript exercise program, taken from UK National Guidance.
  The advice will be directed to be undertaken for 6 weeks immediately prior to surgery.
  Interventions: Behavioral: Exercise Prescription
- Exercise prescription and Virtual Reality Exercise Gaming (Experimental): This group will be provided with a prescript exercise program as in Arm 1. However, this group of patients will also be presented with a Virtual Reality Headset, pre-programmed with Exercise promoted games which will be provided to support and encourage their exercise regimen.
  Again this advice and support will be directed to be undertaken for 6 weeks immediately prior to surgery.
  Interventions: Device: Exercise Prescription and Virtual Reality Exercise Gaming support

INTERVENTIONS:
Behavioral: Exercise Prescription — Standardised Exercise Prescription.
  Arms: Exercise prescription
Device: Exercise Prescription and Virtual Reality Exercise Gaming support — Standardised Exercise Prescription with the additional support of Virtual Reality Promoted Exercise Games.
  Arms: Exercise prescription and Virtual Reality Exercise Gaming

SUMMARY:
Exercise is a vital part of cardiopulmonary conditioning, this means improving general fitness. Undertaking surgery has been likened, physiologically, to running a marathon. It is essential that before any operation the patient undergoing the procedure is as optimised as possible.

Bariatric surgery is no exception. Patients with a high weight often have other conditions most commonly related to the heart and lungs through the excess visceral fat content. This places this group of patients at particular risk of potentially, albeit rare, of having a major and possibly catastrophic cardiac event on the operating table during anaesthetic. Pre-operative conditioning is therefore vital in this group of patients who are often young and not other than their weight necessarily unwell. Exercise plays an important role in the run up to surgery however, many pre-operative exercise prescription programs in the past have failed, often related to the lack of compliance. However, this maybe due to the poor body image they have of themselves presenting in public to the gym or swimming pool.

Current Virtual Reality Games propose that, through their use they encourage exercise and increase heart rate. Given the more personalised nature of this form of media over public engagement, this new media may offer an opportunity to explore whether there is any benefit in terms of pre-conditioning this group of patients prior to their surgery. This study aims, in its first instance, to evaluate whether the Virtual Reality promoted exercise games encourage and can sustain increased activity prior to surgery.

DETAILED DESCRIPTION:
It is estimated that the annual social care costs of obesity to NHS local authorities is £352 million. Obesity surgery currently offers the only long term cure but it carries substantial risk to a group of patients who are often young with other obesity related health concerns; including of the heart and lungs.

The need to improve the condition of the heart and lungs within this patient group prior to surgery is essential. Activity can improve these organs and promote a much lower risk during surgery, reducing the risk of heart attacks or dangerous abnormal rhythms of the heart from occurring during the procedure.

Although exercise alone cannot support long term weight-loss it is vital to promoting a stronger healthier heart in the short term prior to surgery.

This study aims to explore the use of Virtual Reality Gaming to increase activity within this patient group compared to simply encouraging exercise as is undertaken in standard current practice. The initial consideration is as to whether this new media is capable of increasing activity in this group and hopefully improve their heart and lungs going into surgery.

ELIGIBILITY:
Inclusion Criteria:

1. All patients referred to the Weight Management and Obesity Surgery Service at the Royal Cornwall Hospital between January 2020 and December 2020 for Primary Bariatric Surgery.
2. Patients aged 18yrs and over.
3. Patient able to consent (with or without interpreter).
4. Patient able to undergo a general anaesthetic (seen by anaesthetist).

Exclusion Criteria:

1. Patients referred for Revisional Bariatric Surgery.
2. Patients unable to use the Virtual Reality Gaming system.
3. Patient unable to consent.
4. Patients without a clear understanding of the English language.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Activity minutes using Activity tracker | 6 weeks preoperatively
  Measured using Activity tracker
Calories Burnt using Activity Tracker | 6 weeks preoperatively
  Measured using Activity tracker
Heart rate and Heart rate variability using Activity Tracker | 6 weeks preoperatively
  Measured using Activity tracker
Complications at surgery using Clavien-Dindo Classification | 90 days post operatively
  Record of 90 day surgical complications

SECONDARY OUTCOMES:
Total excess Weight-loss post surgery (Kg) | 18 months
  Measurement of weight at postoperative consultations

OTHER OUTCOMES:
Exercise pre-operatively only using Activity Tracker | Each day for 4 weeks prior to surgery
  Measurement of exercise taken

CONTACTS AND LOCATIONS:
Overall Officials: James Clark, FRCS PhD, Principal Investigator — Royal Cornwall Hospitals NHS Trust
Locations (1):
- Royal Cornwall Hospitals Trust, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No